CLINICAL TRIAL: NCT00195143
Title: Phase I Study of Subthalamic GAD Gene Transfer in Medically Refractory Parkinson's Disease Patients
Brief Title: Safety Study of Subthalamic Nucleus Gene Therapy for Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurologix, Inc. (Industry)
Collaborators: Weill Medical College of Cornell University (Other); North Shore University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0902-478
Record Dates: First submitted 2005-09-15; First posted 2005-09-19 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2005-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; GABA; Subthalamic nucleus; Adeno-associated virus; AAV; Gene therapy
MeSH Terms: conditions — Parkinson Disease

INTERVENTIONS:
Genetic: Surgical infusion of AAV-GAD into the subthalamic nucleus

SUMMARY:
The purpose of this study is to determine the safety of using a modified virus to transfer a gene called GAD into a region of the brain called the subthalamic nucleus in patients with advanced Parkinson's disease. The overall goal of this approach is to ultimately normalize the flow of information in several brain regions responsible for movement, to ultimately improve function in patients with this disorder. The current study is primarily designed to evaluate the safety of this approach, but patients are also being monitored for possible signs of effectiveness as well.

DETAILED DESCRIPTION:
This study involves treatment of patients with medically refractory Parkinson's disease (PD) with gene therapy. The patients are chosen from a population of patients who would normally be candidates for standard deep brain stimulation (DBS) surgery for PD. These patients respond to medical therapy, but develop substantially reduced responses over time, often with severe fluctuations in their condition between a functional and severely non-functional state. Some patients also develop dose-limiting side effects from medication, including involuntary movements called dyskinesias and nightmares. When there are no medical contraindications, DBS is often performed in these patients to try to quiet hyperactive brain regions such as the subthalamic nucleus (STN). In PD, the STN is overactive due to a loss of GABA inputs to this region, which normally reduces neuronal firing. In turn, the STN drives other brain regions, including the globus pallidus (GPi) and substantia nigra (SNr), which are also hyperactive and which also have reduced GABA inputs. The goal of this gene therapy trial is to introduce the gene for glutamic acid decarboxylase (GAD) into the STN using an adeno-associated virus (AAV) vector, in order to permit the STN to produce it's own GABA, as well as release GABA into the GPi and SNr targets, which also have reduced GABA inputs. This is anticipated to restore a more normal pattern of information flow from this basal ganglia circuit to the thalamus and higher cortical structures in order to reduce the motor symptoms of PD, while eliminating complications arising from inserting DBS electrodes and batteries into the human body.

ELIGIBILITY:
Inclusion Criteria:

* Duration of disease: Greater than 5 years
* Idiopathic Parkinson's disease
* Parkinson's medication stable for 3 months
* Absence of dementia
* Hoehn and Yahr rating: 3 or greater and/or UPDRS: 30 or more in "off" state and/or Complications of l-dopa therapy limiting effective use

Exclusion Criteria:

* Poor candidate for any surgery
* Significant dementia
* Secondary parkinsonism
* Severe autonomic symptoms
* Atypical Parkinson's disease
* History of substance abuse

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2003-08; Study Completion 2005-08

PRIMARY OUTCOMES:
Safety

SECONDARY OUTCOMES:
Improvement in brain metabolism measured by PET scans
Improvement in standard clinical rating scales

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Kaplitt, MD PhD, Principal Investigator — Weill Medical College of Cornell University; Matthew J During, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

REFERENCES:
- [Background] Luo J, Kaplitt MG, Fitzsimons HL, Zuzga DS, Liu Y, Oshinsky ML, During MJ. Subthalamic GAD gene therapy in a Parkinson's disease rat model. Science. 2002 Oct 11;298(5592):425-9. doi: 10.1126/science.1074549. PMID 12376704
- [Derived] Kaplitt MG, Feigin A, Tang C, Fitzsimons HL, Mattis P, Lawlor PA, Bland RJ, Young D, Strybing K, Eidelberg D, During MJ. Safety and tolerability of gene therapy with an adeno-associated virus (AAV) borne GAD gene for Parkinson's disease: an open label, phase I trial. Lancet. 2007 Jun 23;369(9579):2097-105. doi: 10.1016/S0140-6736(07)60982-9. PMID 17586305